CLINICAL TRIAL: NCT02872779
Title: Correlation Between Circulating Tumour Markers Early Variations and Clinical Response in First Line Treatment of Metastatic Colorectal Cancer
Acronym: COCA-MACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Diagnostic
Other Study IDs: 2015/076/HP
Record Dates: First submitted 2016-08-16; First posted 2016-08-19 (Estimated); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Circulating Markers; Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients Treated for Metastatic Colorectal cancer (Experimental): Blood sampling for free mutant DNA analysis for Patients Treated for Metastatic Colorectal cancer
  Interventions: Procedure: Blood sampling for free mutant DNA analysis

INTERVENTIONS:
Procedure: Blood sampling for free mutant DNA analysis — Blood sampling for Patients Treated for Metastatic Colorectal cancer

SUMMARY:
The chemotherapy monitoring is currently based on radiological (RECIST 1.1 guideline) and clinical evaluation every 3 months. Circulating markers as Carcino Embryonic Antigen (CEA), circulating tumour DNA and total cell free DNA represent an alternative approach to evaluate the response. In the field of metastatic colorectal cancer (mCRC) recent studies suggest that early evaluation could be clinically relevant. Indeed, early tumoral response seems to be correlated to overall survival. Moreover, post-operative morbidity increases with the number of prior chemotherapy treatments. Early evaluation could allow to modify chemotherapy regimens when response appears to be insufficient.

The aim of the present study is to evaluate, in a prospective cohort of patients treated with systemic IV chemotherapy (5 Fluorouracil +/- oxaliplatin +/- irinotecan) +/- targeted therapy as first line treatment for a mCRC, the correlation between early variations of circulating tumour markers including CEA, circulating tumour DNA and total cell free DNA, and the 3 months objective response as defined in the RECIST 1.1 guideline.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age superior to 18 years.
* Histologically confirmed metastatic colorectal adenocarcinoma.
* Measurable disease according to the RECIST 1.1 guideline
* ECOG performance status <3.
* Disease requiring IV chemotherapy (5 Fluorouracil +/- oxaliplatin +/- irinotecan) +/- targeted therapy (cetuximab or panitumumab or bevacizumab) every 14 days
* No prior chemotherapy for this adenocarcinoma with the exception of adjuvant chemotherapy
* Signed and dated informed consent document.

Exclusion Criteria:

* Medical history of cancer within 5 years
* Medical contraindication for a treatment consisted of IV chemotherapy (5 Fluorouracil +/- oxaliplatin +/- irinotecan) +/- targeted therapy (cetuximab or panitumumab or bevacizumab)
* Patient with known psychiatric or substance abuse disorders that could interfere with cooperation with the requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2016-07-18 (Actual); Primary Completion 2020-08-10 (Actual); Study Completion 2020-08-10 (Actual)

PRIMARY OUTCOMES:
Difference from baseline in the number of free mutant DNA in blood | 5 weeks
  Variation of free mutant DNA kinetic at week 5 to predict tumor progression at 3 months (Evaluation based on the RECIST 1.1 guideline)

SECONDARY OUTCOMES:
Difference from baseline in the number of free mutant DNA in blood | 3 weeks
  Variation of free mutant DNA kinetic at week 3 to predict tumor progression at 3 months (Evaluation based on the RECIST 1.1 guideline)
Evaluation of response based on the RECIST 1.1 guideline | 3 Months
  sensitivity and specificity of free mutant DNA kinetic at Week 5 (RECIST) to predict tumor progression at 3 months (RECIST)

CONTACTS AND LOCATIONS:
Overall Officials: Alice GANGLOFF, MD, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: Undecided